CLINICAL TRIAL: NCT06388200
Title: A Phase 3, Multi-Center, Randomized Study to Assess The Efficacy, Safety and Tolerability of Subretinal OCU400 Gene Therapy for the Treatment of Retinitis Pigmentosa
Brief Title: A Phase 3 Study Of OCU400 Gene Therapy for the Treatment Of Retinitis Pigmentosa
Acronym: liMeliGhT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCU400-301
Record Dates: First submitted 2024-04-09; First posted 2024-04-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa
Keywords: Modified Gene therapy; Retinitis Pigmentosa; RHO; RP; NR2E3; Subretinal Injection
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is outcome assessor blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RHO Arm (Experimental): Subjects will receive a sub-retinal injection of OCU400-301 modifier gene therapy product with a concentration of 2.5 x 10^10 vg/eye
  Interventions: Genetic: Sub-Retinal Administration of OCU400-301
- Gene Agnostic Arm (Experimental): Subjects will receive a sub-retinal injection of OCU400-301 modifier gene therapy product with a concentration of 2.5 x 10^10 vg/eye
  Interventions: Genetic: Sub-Retinal Administration of OCU400-301
- Control for RHO Arm (No Intervention): Will not receive any active study intervention
- Control for Gene Agnostic Arm (No Intervention): Will not receive any active study intervention

INTERVENTIONS:
Genetic: Sub-Retinal Administration of OCU400-301 — Sub-Retinal Administration of OCU400-301
  Arms: Gene Agnostic Arm; RHO Arm

SUMMARY:
This is a Phase 3 study to Assess the Efficacy, Safety and Tolerability of OCU400 in patients with retinitis pigmentosa (RP) associated with RHO mutations and patients with any other RP associated mutation with a clinical phenotype of RP.

This is a multicenter, assessor blinded and randomized study which will enroll 150 subjects.

DETAILED DESCRIPTION:
A total of one hundred and fifty (150) RP participants will be enrolled in this study- 75 in each of either two arms, RHO arm (n=75) or Gene agnostic arm (n=75). RHO arm will only enroll participants with confirmed genetic diagnosis of mutation in RHO gene; whereas Gene Agnostic arm will enroll RP Participants based on clinical diagnosis of RP and a confirmed genetic diagnosis with a gene associated with RP.

Subjects in each arm will be randomized into treatment (N=50) and control groups (N=25). Subjects in the treatment group will receive a sequential, bilateral sub-retinal injection of OCU400 if both eyes meet inclusion criteria. Control or untreated group subjects will receive OCU400 subretinal injection after completion of 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 3 years of age
2. Confirmed genetic diagnosis of autosomal dominant RHO mutation with clinical diagnosis of RP
3. Clinical Diagnosis of Syndromic or Non-Syndromic RP with/without confirmed genetic diagnosis of any other RP associated mutation (except AD-NR2E3)
4. BCVA ≤ 80 letters and ≥25 letters as measured by an ETDRS chart
5. Visual field of >5° in any meridian as measured by a III4e isopter or equivalent
6. Able to perform a Luminance LDNA at certain light intensity at the Screening visit
7. Presence of photoreceptors as determined by SD-OCT

Exclusion Criteria:

1. Subject lacks evidence of outer nuclear layer
2. Previous treatment with a gene-therapy or cell therapy product or treatment with any investigational drug or ocular device within one year.
3. History of any corticosteroid contraindication, corticosteroid related IOP spikes or uncontrolled glaucoma.
4. Cataract surgery within 3 months. YAG capsulotomy within 1 month. Any other intraocular surgery within 6 months.
5. Active ocular/intraocular infection, any history of rhegmatogenous retinal detachment or Current retinal detachment or retinal implant.
6. Breast-feeding, pregnancy, sperm donation or inability to practice strict contraception

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with change in functional vision in the study eye of RP subjects as assessed by LDNA | 52 weeks
  Change in the LDNA assessment from screening in the study eye of RP subjects with RHO mutation will be compared to controls
Number of participants with change in functional vision in the study eye in Gene Agnostic group as assessed by LDNA | 52 weeks
  Change in the LDNA assessment from screening in the study eye in Gene Agnostic Arm subjects will be compared to controls

SECONDARY OUTCOMES:
Number of participants with change in functional vision in the all treated eyes of RP subjects as assessed by LDNA | 52 weeks
  Change in the LDNA assessment from screening in all treated eyes of RP subjects with RHO mutation will be compared to controls
Number of participants with change in functional vision in the all treated eyes of subjects in Gene Agnostic Arm as assessed by LDNA | 52 weeks
  Change in the LDNA assessment from screening in all treated eyes of subjects in Gene Agnostic Arm subjects will be compared to controls
Number of participants with change in visual function in subjects with RHO mutation as assessed by LLVA letter score | 52 weeks
  Change in LLVA letter scores in RP subjects with mutations in RHO will be compared to controls
Number of participants with change in visual function in Gene Agnostic Arm as assessed by LLVA letter scores | 52 weeks
  Change in LLVA letter scores in Gene Agnostic Arm subjects will be compared to controls
Ocular and non-ocular Events | 52 weeks
  Incidence and severity of Study Drug-related adverse events (SDAE), Treatment-Emergent adverse events (TEAEs), Serious adverse events (SAEs) and Adverse Events of Special Interest (AESI).

OTHER OUTCOMES:
Patients Global Impression of Change (PGIC) score | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qamar, Study Chair — Ocugen
Locations (17):
- United States (12):
  - Associated Retina Consultants, Phoenix, Arizona
  - University of Southern Califormia, La Jolla, California
  - University of Southern California, Roski Eye Insitute, Los Angeles, California
  - Advanced Research, LLC., Deerfield Beach, Florida
  - Bascom Palmer Eye Institute, University of Miami, Miller School of Medicine, Miami, Florida
  - Erie Retina Research LLC, Erie, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Gundersen Health System, La Crosse, Wisconsin
- Canada (5):
  - Calgary Retina Consultants, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - The University of British Columbia, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No